CLINICAL TRIAL: NCT03257774
Title: A Pilot Evaluation of Newly Developed Adhesives and How They Are Impacted by Output
Brief Title: Evaluation of the Effect of Output on New Adhesives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP265_12_13_14
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test of three new adhesive strips (Experimental): The subjects test three new adhesive strips
  * adhesive strip A
  * adhesive strip B
  * adhesive strip C
  Interventions: Other: Adhesive strip A; Other: Adhesive strip B; Other: Adhesive strip C

INTERVENTIONS:
Other: Adhesive strip A — Strip consisting of a newly developed adhesive
Other: Adhesive strip B — Strip consisting of a newly developed adhesive
Other: Adhesive strip C — Strip consisting of a newly developed adhesive

SUMMARY:
The study investigates the impanct real output has on the adhesion of a new adhesive

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Have had a stoma for more than one year
4. Have intact skin on the area used in the evalua-tion
5. Has a stoma with a diameter up to (≤) 35 mm
6. Have a peristomal area accessible for application of adhesive strips (assessed by investigating scientist)

Exclusion Criteria:

1. Currently receiving or have within the past 2 month received radio- and/or chemotherapy
2. Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment.
3. Are pregnant or breastfeeding
4. Having dermatological problems in the peristo-mal- or abdominal area (assessed by investigating scientist)
5. Actively participating in other interventional clinical investigations or have previously participated in this investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2017-09-13 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
Trans epidermal water loss | 8 hours
  The trans epidermal water loss is measured on the peristomal skin using a probe. Thrans epidermal water loss is a measure for the skins barrier function. There is always a loss of water from the skin du to natural evaporation. However, when the skin barrier is damaged more water can evaporate. Trans epridermal water loss is used to assess the damage to the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Nielsen, Principal Investigator — Head of preclinical department
Locations (1):
- Coloplast A/S, Humlebæk, Denmark